CLINICAL TRIAL: NCT06154096
Title: Response to Glucagon in Patients With Metabolic-associated Steatotic Liver Disease: a Feasibility Study
Brief Title: Liver Fat and Glucagon Resistance
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 334557
Record Dates: First submitted 2023-11-15; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Steatosis of Liver
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, faeces, urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy volunteer: Subject without MASLD or metabolic-associated disease
  Interventions: Other: Acute glucagon infusion
- MASLD: Subject with MASLD
  Interventions: Other: Acute glucagon infusion

INTERVENTIONS:
Other: Acute glucagon infusion — All subjects will undergo an amino acid infusion and pancreatic clamp during which they will have stable isotope turnover of glucose and alanine measured in two steady state periods - firstly, with low-dose glucagon infusion and secondly, with high-dose glucagon infusion

SUMMARY:
One in four adults worldwide have too much fat stored in the liver which is known as metabolic associated steatotic liver disease (MASLD). This was previously known as non- alcoholic fatty liver disease (NAFLD). This can lead to liver failure and death in severe cases. Unfortunately, there are no specific drugs to treat MASLD.

Glucagon is a natural hormone that controls how the body stores and uses fuel. Glucagon acts on liver cells to use protein and fat to make sugar. It decreases the amount of liver fat.

The investigators think that patients with MASLD may not respond to the actions of glucagon. This could contribute to the build-up of fat in the liver.

In this study the investigators will be investigating the effects of glucagon on protein breakdown and sugar production in patients with and without MASLD.

Healthy volunteers and patients with MASLD will attend for one study visit each which will last for 4-5 hours. During this time they will have infusions into a vein of glucagon and other hormones, amino acids (to mimic the fed state) and 'tracers'. From another vein they will have several blood samples during this period. By analysing these blood samples the investigators will be able to measure the effects of glucagon on protein and glucose turnover (metabolism), and whether this differs between healthy volunteers and those with MASLD.

If the investigators find that patients with MASLD are resistant to the actions of glucagon, this could help with the development of drugs to treat MASLD.

DETAILED DESCRIPTION:
This is a feasibility cohort-control experimental medicine study. Participants will attend for one study visit lasting 4-5 hours. The study will involve a maximum of 10 healthy volunteers and 10 patients with MASLD. All subjects will undergo an amino acid infusion and pancreatic clamp during which they will have stable isotope turnover of glucose and alanine measured in two steady state periods - firstly, with low-dose glucagon infusion and secondly, with high-dose glucagon infusion. The studies will take place in the Clinical Research Unit at Hammersmith Hospital, Imperial College.

Screening visit:

During this visit that will last around an hour, prospective participants will have a consultation with a study doctor. The doctor will assess medical history and explain the study. They will also perform a routine physical examination and take some blood tests. Women of child-bearing age will undergo urinalysis to exclude pregnancy. Participants will be contacted a couple of days later to let discuss blood test results, and if these are satisfactory they will be invited to attend for 1 study visit.

Study visit:

Participants will be asked to avoid alcohol and strenuous exercise for 24 hours before the study visit. They will be asked to fast (that is, consume nothing except water) for 10-14 hours before the visit. The visits will start at around 8 or 9am and finish at about 1 or 2pm.

On arrival, female volunteers will be asked for a urine specimen which will be tested for evidence of pregnancy. Participants will be weighed and have pulse, blood pressure and temperature checked.

The participant's arms will be loosely wrapped in a heating pad (50°C). A study investigator will insert two cannulae (thin flexible tubes) into a vein in each arm. One cannula will be used for infusions and the other for blood samples. The investigators will infuse glucagon and two other hormones (insulin and somatostatin), amino acids (to mimic the 'fed state') and 'tracers' of an amino acid called alanine and glucose. The investigators will take multiple blood samples at intervals during the infusions to measure the levels of hormones, sugar and protein in the blood. The total amount will be less than 200ml (around 11 tablespoons), which is less than half the amount taken during a blood donation session.

After 3.5 hours the cannulae will be removed, the participant will be offered something to eat, and after 15-30 minutes of observation they will be allowed to leave the unit. During the study participants can watch TV or read. They will not be able to eat but they can sip water.

ELIGIBILITY:
INCLUSION CRITERIA (all patients)

* Male or female
* Able to give full informed consent
* 18 years old or more (children have different metabolism)

INCLUSION CRITERIA (healthy volunteers) • Normal FIB4 (<1.3; this indicates no evidence of liver fibrosis)

INCLUSION CRITERIA (patients with MASLD)

• Biopsy-proven or clinically diagnosed MASLD (>5% steatosis)

EXCLUSION CRITERIA (all patients)

* Current or history of any medical condition that could interfere with the study or potentially cause harm to the participant
* Pregnant or breastfeeding (affects metabolism)
* Recent weight loss or gain (>10% in previous 3 months)
* History of hypersensitivity to any of the infusates listed in the study design
* Diabetes or pre-diabetes (HbA1C >42mmol/mol)
* Consumption of over 14 units of alcohol per week

EXCLUSION CRITERIA (healthy volunteers)

* Evidence of metabolic syndrome
* Previous or current clinical or biochemical evidence of liver disease

EXCLUSION CRITERIA (patients with MASLD)

* Evidence of liver cirrhosis
* Non-metabolic associated causes of liver disease (e.g. viral hepatitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and patients with MASLD
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Standard deviation of alanine turnover | one study visit = 1 day per volunteer, 20 study visits, 3 months in total
  Standard deviation of differences in alanine turnover between two steady state periods (low and high dose glucagon infusion) for use in a subsequent sample size calculation
Standard deviation of glucose turnover | one study visit = 1 day per volunteer, 20 study visits, 3 months in total
  Standard deviation of differences in glucose turnover between two steady state periods (low and high dose glucagon infusion) for use in a subsequent sample size calculation

SECONDARY OUTCOMES:
Plasma glucagon | one study visit = 1 day per volunteer, 20 study visits, 3 months in total
  Differences in plasma glucagon between two steady state periods (low and high dose glucagon infusion) insulin, lactate, free fatty acids, total amino acids and urea between two steady state periods (low and high dose glucagon infusion)
Plasma insulin | one study visit = 1 day per volunteer, 20 study visits, 3 months in total
  Differences in plasma insulin between two steady state periods (low and high dose glucagon infusion) insulin, lactate, free fatty acids, total amino acids and urea between two steady state periods (low and high dose glucagon infusion)
Plasma lactate | one study visit = 1 day per volunteer, 20 study visits, 3 months in total
  Differences in plasma lactate between two steady state periods (low and high dose glucagon infusion) insulin, lactate, free fatty acids, total amino acids and urea between two steady state periods (low and high dose glucagon infusion)
Plasma free fatty acids | one study visit = 1 day per volunteer, 20 study visits, 3 months in total
  Differences in plasma free fatty acids between two steady state periods (low and high dose glucagon infusion) insulin, lactate, free fatty acids, total amino acids and urea between two steady state periods (low and high dose glucagon infusion)
Plasma total amino acids | one study visit = 1 day per volunteer, 20 study visits, 3 months in total
  Differences in plasma total amino acids between two steady state periods (low and high dose glucagon infusion) insulin, lactate, free fatty acids, total amino acids and urea between two steady state periods (low and high dose glucagon infusion)
Plasma urea | one study visit = 1 day per volunteer, 20 study visits, 3 months in total
  Differences in plasma urea between two steady state periods (low and high dose glucagon infusion) insulin, lactate, free fatty acids, total amino acids and urea between two steady state periods (low and high dose glucagon infusion)
Plasma metabolite composition | one study visit = 1 day per volunteer, 20 study visits, 3 months in total
Urine metabolite composition | one study visit = 1 day per volunteer, 20 study visits, 3 months in total
Plasma lipid composition | one study visit = 1 day per volunteer, 20 study visits, 3 months in total
Urine lipid composition | one study visit = 1 day per volunteer, 20 study visits, 3 months in total
Microbiome composition of stool | one study visit = 1 day per volunteer, 20 study visits, 3 months in total
  Method: sequencing of 16S rRNA

CONTACTS AND LOCATIONS:
Overall Officials: Emma Rose McGlone, PhD, Principal Investigator — Imperial College London

IPD SHARING:
Plan to Share IPD: No